CLINICAL TRIAL: NCT00742391
Title: A Multi-center, Randomized, Parallel Group, Double-blind, Vehicle-controlled Study to Evaluate the Efficacy and Safety of PEP005 (Ingenol Mebutate) Gel, 0.05% In Patients With Actinic Keratoses ON Non-head Locations (REGION-I)
Brief Title: A Multicenter Study to Evaluate the Efficacy and Safety of PEP005 (Ingenol Mebutate) Gel When Used to Treat Actinic Keratoses (AKs) on the Non Head Locations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEP005-014
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2012-03-21 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Actinic Keratoses
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): PEP005 (ingenol mebutate) Gel
  Interventions: Drug: PEP005 (ingenol mebutate) Gel
- 2 (Placebo Comparator): Vehicle gel
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: PEP005 (ingenol mebutate) Gel — two day treatment
  Arms: 1
Drug: Vehicle gel — two day treatment
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether topical application of PEP005 is effective for the treatment of actinic keratoses.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age.
* Female patients must be of:
* Non-childbearing potential;
* Childbearing potential, provided negative serum and urine pregnancy test and using effective contraception.
* 4 to 8 AK lesions on non-head locations.

Exclusion Criteria:

* Cosmetic or therapeutic procedures within 2 weeks and within 2 cm of the selected treatment area.
* Treatment with immunomodulators, or interferon/ interferon inducers or systemic medications that suppress the immune system within 4 weeks.
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy within 8 weeks and 2 cm of treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (18):
  - Omni Dermatology Research, Mesa, Arizona
  - Colorado Medical Research Center, Denver, Colorado
  - Advanced Dermatology and Cosmetic Research, Kissimmee, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Advanced Dermatology & Cosmetic Surgery, Ormond Beach, Florida
  - Medaphase Inc, Newnan, Georgia
  - Gwinnett Clinical Research Centre, Snellville, Georgia
  - Dermatology Center of Indiana/Indiana Clinical Trials Center, Plainfield, Indiana
  - Henry Ford Health Systems, Detroit, Michigan
  - Karen S. Harkaway, MD. LLC, South Delran, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Associates of Rochester, Rochester, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon Medical Research, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Dermatology East, Germantown, Tennessee
  - Rivergate Dermatology and Skin Care Center, Goodlettsville, Tennessee
  - J & S Studies, Inc., College Station, Texas
- Australia (2):
  - The Skin Centre, Benowa, Queensland
  - Burswood Dermatology, Victoria Park, Western Australia

REFERENCES:
- [Derived] Lebwohl M, Swanson N, Anderson LL, Melgaard A, Xu Z, Berman B. Ingenol mebutate gel for actinic keratosis. N Engl J Med. 2012 Mar 15;366(11):1010-9. doi: 10.1056/NEJMoa1111170. PMID 22417254
- See also: Food and Drug Authority — http://www.fda.gov/
- See also: Therapeutic Goods Administration — http://www.tga.gov.au/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period was 05 September 2008 (first patient randomized) to 23 February 2009 (last patient completed Day 57)
Groups:
- PEP005 (Ingenol Mebutate) Gel: PEP005 (ingenol mebutate) Gel 0.05% once daily for 2 consecutive days
- Vehicle Gel: Vehicle gel once daily for 2 consecutive days
Period: Overall Study
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Started | 126 | 129
Completed | 122 | 128
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel | Total
Number analyzed (Participants) | 126 | 129 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.59) | 66.9 (9.89) | 67.1 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 56 | 96
  Male | 86 | 73 | 159
Region of Enrollment [Number; unit: participants]
  United States | 110 | 116 | 226
  Australia | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Patients With Complete Clearance of Actinic Keratosis (AKs)
Description: Complete clearance rate of actinic keratosis (AK) lesions defined as the proportion of patients with no clinically visible AK lesions in the selected treatment area.
Time Frame: 57 days
Population: Intention to treat population
Measure: Number; unit: Participants
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Number analyzed (Participants) | 126 | 129
Participants | 35 | 6
Statistical Analysis 1: Comparison: PEP005 (Ingenol Mebutate) Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Patients With Partial Clearance of Actinic Keratosis (AKs)
Description: Partial clearance rate of AK lesions defined as the proportion of patients with a 75% or greater reduction in the number of actinic keratosis (AK) lesions identified at baseline in the selected treatment area.
Time Frame: baseline and 57 days
Population: Intention to treat population
Measure: Number; unit: participants
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Number analyzed (Participants) | 126 | 129
participants | 56 | 6
Statistical Analysis 1: Comparison: PEP005 (Ingenol Mebutate) Gel vs Vehicle Gel; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 57 days
Description: One patient in the PEP005 Gel, 0.05% group discontinued study medication (Day 2 dose not applied) due to an AE (application site pain)
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 1/125 | 3/129
Other Adverse Events (participants affected / at risk) | 0/125 | 0/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEP005 (Ingenol Mebutate) Gel (N=125) | Vehicle Gel (N=129)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Lymphoma (neck) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the Study is completed, Institution shall have the right to publish their own data resulting from the Study upon the earlier of (a) publication of a multi-center publication coordinated by Sponsor or (b) the date of submission of the data resulting from the Study by Sponsor to the FDA. Institution shall furnish Sponsor with a copy of any proposed publication or release at least 90 days in advance of the proposed submission or presentation date.